CLINICAL TRIAL: NCT01856049
Title: Umbilical Cord Blood Collection and Processing for Severe Congenital Heart Disease
Brief Title: Umbilical Cord Blood Collection and Processing for Hypoplastic Left Heart Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Susana Cantero Peral, M.D., Ph.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-007176
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Hypoplastic Left Heart Syndrome (HLHS)
Keywords: HLHS; Hypoplastic Left Heart Syndrome; UCB (umbilical cord blood); Umbilical cord blood; Cord blood; Cardiac regeneration
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbilical Cord Blood Collection (Other): Umbilical Cord Blood is drawn from the umbilical cord of newborn babies diagnosed with Hypoplastic Left Heart Syndrome, before placental detachment. Cord blood is packaged in a Credo Cube, and sent at a temperate state to the manufacturer immediately after draw. At least 65 mL of cord blood is needed to produce a stem cell product during manufacturing. Once processed, the patient's autologous cord blood stem cells will be frozen for their potential future use in a clinical trial.
  Interventions: Other: Collection of umbilical cord blood

INTERVENTIONS:
Other: Collection of umbilical cord blood — Cord blood will be processed in the temperate state it was collected to produce a pure, stem cell product identifiable to patients with Hypoplastic Left Heart Syndrome, and will be stored at a frozen state for their potential, future use in a clinical trial.

SUMMARY:
Cell-based cardiac regeneration has been the focus of acquired, adult heart disease for many years. However, congenital heart disease with severe structural abnormalities may also be reasonable targets for cell-based therapies. Interestingly, the pediatric heart is naturally growing and may be the most amendable to regenerative strategies. Therefore, identifying autologous cells (cells from the patient's own body) would be important to initiate these studies.

This study aims to validate the use of umbilical cord blood as a source of autologous cells for the purpose of cardiac repair of congenital heart disease. Cells will be isolated from the cord blood to help us determine the feasibility of collection, processing, and storage of these samples at the time of birth of infants with prenatal diagnosis of hypoplastic left heart syndrome. This study may be useful for the development of pre-clinical and clinical studies aimed at the long-term goal of repairing damaged heart muscle.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is an abnormal formation that occurs during the development of a baby's heart, heart valves and/or large vessels such as the aorta artery. CHD is the most common cause of major congenital defects accounting for almost 30% of all defects. While the statistics vary among studies, the best birth prevalence estimate is 8 per 1000 live births. In the USA, CHD affects 1% of all births per year, with an estimated 40,000 babies born with any type of heart defect every year.

The important improvements in CHD diagnosis and surgical treatment in the last decades has led to an increased survival of newborns affected with heart defects. A large number of CHD can be diagnosed during pregnancy, and the patients can present a broad range of symptoms. Forms of CHD are usually classified based on their severity, from mild to severe. One of the mildest forms of CHD is atrial septal defect, which can be undetectable until adulthood and VSD. On the other hand, severe CHD that requires multiple palliative surgeries includes single ventricle defects, such as hypoplastic left heart syndrome (HLHS), and tricuspid atresia.

The survival of infants with CHD will depend on the severity of the defect and the time of diagnosis and treatment received. The one-year survival of newborns with severe or critical CHD (generally any type of surgery/procedures in their first year of life) is estimated to be 75%.

Stem cell therapy has emerged as a new paradigm of treatment in the field of CHD with promising results. Cardiac regeneration has been the focus of acquired, adult heart disease for many years. However, congenital heart disease with structural abnormalities may also be a good target for other research studies. In fact, the pediatric heart is naturally growing and may be amendable to regenerative strategies. Furthermore, the initial pre-clinical and clinical studies have demonstrated that the delivery of stem cells into the heart of patients with CHD is feasible and safe. Moreover, the cell therapy approach, along with the standard surgical palliation, seems to offer benefits over surgical treatment alone. Even though the number of cell therapy clinical trials for CHD has increased in the last decade, more long-term follow-up studies are needed in this population setting in order to define the role of stem cell therapy in the clinical practice. Therefore, confirming our ability to produce autologous cells (cells from the patient's own body) from patients with severe CHD is an important step towards the long-term goal of being able to discover innovative cell-based protocols.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman, regardless of age, with a prenatal diagnosis of severe CHD/hypoplastic left heart syndrome.
* One or both parents willing to consent to the storage of umbilical cord blood for the specific purpose of regenerative research
* Delivering party and/or expectant family is willing to sign Release of Information to request fetal echo text report diagnosing severe CHD/hypoplastic left heart syndrome
* Parent(s) willing to be contacted 60 days after collection for follow-up screening questions regarding the health status of the baby affected with severe CHD/hypoplastic left heart syndrome.

Exclusion Criteria:

* Individuals unwilling to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2012-05; Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Percent of samples contaminated | 14 days after collection
Percent of cells that are viable following post thaw analysis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Susana Cantero Peral, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials